CLINICAL TRIAL: NCT01829035
Title: A Randomized, Controlled Phase III Trial of Sorafenib With or Without Conventional Transarterial Chemoembolization in Patients With Advanced Hepatocellular Carcinoma (STAH Study)
Brief Title: A Randomized, Controlled Phase III Trial of Sorafenib With or Without cTACE in Patients With Advanced HCC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Joong-Won Park, Chief of Hepatology, Center for Liver Cancer, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STAH Korea Trial
Record Dates: First submitted 2013-03-31; First posted 2013-04-11 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Advanced Adult Hepatocellular Carcinoma
Keywords: TACE; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm S (No Intervention): sorafenib 400mg bid daily po until progression
- Arm C (Experimental): after the first Conventional Transarterial Chemoembolization is completed, sorafenib po and cTACE on demand until progression
  Interventions: Other: Conventional Transarterial Chemoembolization (cTACE)

INTERVENTIONS:
Other: Conventional Transarterial Chemoembolization (cTACE) — Concurrent use of the following material/drug is defined as cTACE in this trial.
  * Embolization material (e.g., gelatin sponges, porous gelatin particles, Ivalon, etc.) other than ethiodized oil
  * Anti-tumor drug:
    1. Unapproved drug/embolization material from each regulatory agency should not be used.
    2. To chemo-embolize all arteries feeding viable lesions via super selective cTACE, which is more effective and can be recommended as it rarely causes impairment of non-cancerous liver tissues. After assessing the disappearance of tumor stain as much as possible by angiography, the cTACE procedure should be completed
  Arms: Arm C

SUMMARY:
This is a randomized, multi-center, open-labeled, phase III study in patients with advanced HCC. A total of 338 patients will be randomized (1:1) into one of the two treatment arms, to receive sorafenib with (Arm Combination-treatment; Arm C) or without (Arm Sorafenib alone treatment; Arm S) cTACE.

All the patients will be initially given sorafenib within 72 hours after the randomization. Treatment should continue until the criteria for treatment discontinuation are met.

After the treatment period, patients will undergo follow up for survival every 12 weeks (±7 days) from the last dose, and the survival follow up will be performed for at least 1.5 years after the last patient's last treatment.

DETAILED DESCRIPTION:
The superiority of the Arm C (cTACE+Sorafenib) over the Arm S (Sorafenib) in the OS period will be verified in the ITT set and FAS using a stratified log-rank test. Stratification factors consist of mUICC stage (III vs. IV), Vascular invasion (none and Vp1-2 vs. Vp3-4 and any other presence), Child-Pugh score (5 vs. 6-7), serum AFP level (≥200 ng/mL vs. <200 ng/mL). The significance level is 5% (one-sided).

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in the study, patients must meet the following criteria:

1. Signed written informed consent
2. Clinical or histological diagnosis of HCC based on the guidelines of the Korean Liver Cancer Study Group and the National Cancer Center Korea
3. At least one typical enhanced index lesion in the liver that is bi-dimensionally measurable by multiphasic spiral CT scan or dynamic contrast-enhanced MRI, and size of largest tumor is 15 cm or less at enrollment.
4. Tumor conditions confirmed by abdominal imaging (contrast enhanced CT ± MRI) and chest imaging (CT) performed within 4 weeks prior to the treatment initiation:
5. Age of at least 20 years.
6. ECOG Performance Status of 0, 1 or 2.
7. Child-Pugh class A or B (Child-Pugh score ≤ 7).
8. Life expectancy of at least 16 weeks.
9. Adequate bone marrow, liver, and renal function as assessed by the following laboratory requirements (no transfusion, no restoration), conducted within 14 days prior to screening:
10. Female patients at least 1 year postmenopausal, surgically sterile or those of childbearing potential must have a negative urine pregnancy test within 14 days prior to the first treatment, and have to use at least one medically acceptable and effective contraceptive method for the last 2 months prior to Screening Visit: methods of effective contraception result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as a barrier method (implant, injectable contraceptives, oral contraceptives, intrauterine contraceptive device), hormonal IUD, sexual abstinence or vasectomized partner.

Exclusion Criteria:

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Actual)
Dates: Start 2013-02-21 (Actual); Primary Completion 2017-06-21 (Actual); Study Completion 2017-06-21 (Actual)

PRIMARY OUTCOMES:
The overall survival (OS) of oral sorafenib given as monotherapy daily compared to sorafenib with combination cTACE in subjects | 3.5 years

SECONDARY OUTCOMES:
Time to progression (TTP)in patients | 3.5 years
Tumor response rate (TRR)in patients | 3.5 years
Progression free survival(PFS)will be evaluated | 3.5 years
Evaluation of adverse events | 3.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Joong-Won Parkr, Ph.D., Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Korea, Seoul, South Korea

REFERENCES:
- [Derived] Park JW, Kim YJ, Kim DY, Bae SH, Paik SW, Lee YJ, Kim HY, Lee HC, Han SY, Cheong JY, Kwon OS, Yeon JE, Kim BH, Hwang J. Sorafenib with or without concurrent transarterial chemoembolization in patients with advanced hepatocellular carcinoma: The phase III STAH trial. J Hepatol. 2019 Apr;70(4):684-691. doi: 10.1016/j.jhep.2018.11.029. Epub 2018 Dec 6. PMID 30529387